CLINICAL TRIAL: NCT01791972
Title: A Single-Dose Study to Assess the Efficacy of Albuterol SPIROMAX® in Adult and Adolescent Patients With Exercise-Induced Bronchoconstriction (EIB)
Brief Title: Efficacy of Albuterol SPIROMAX® in Adult and Adolescent Patients With Exercise-Induced Bronchoconstriction (EIB)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABS-AS-302
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Results first posted 2015-05-19 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-05

CONDITIONS: Exercise-Induced Bronchoconstriction (EIB)
Keywords: Exercise-Induced Bronchoconstriction (EIB); Spiromax®; Albuterol sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albuterol Spiromax / Placebo Spiromax (Experimental): Albuterol Spiromax, 180 mcg (2 inhalations of 90 mcg/inhalation), single dose on Day 1. Placebo Spiromax (2 inhalations), single dose on approximately Day 7.
  Interventions: Drug: Albuterol Spiromax; Drug: Placebo Spiromax
- Placebo Spiromax / Albuterol Spiromax (Experimental): Placebo Spiromax, (2 inhalations), single dose on Day 1. Albuterol Spiromax 180 mcg (2 inhalations of 90 mcg/inhalation), single dose on approximately Day 7.
  Interventions: Drug: Albuterol Spiromax; Drug: Placebo Spiromax

INTERVENTIONS:
Drug: Albuterol Spiromax — Albuterol Spiromax is an inhalation-driven, multi-dose dry powder inhaler (DPI) containing a blend of albuterol sulfate with alpha-lactose monohydrate. Each actuation represents a dose of 90 mcg of albuterol sulfate. Participants received one dose of two inhalations (180 mcg).
  Other Names: Albuterol DPI, ProAir® RespiClick
Drug: Placebo Spiromax — Placebo Spiromax is an inhalation-driven, multi-dose dry powder inhaler (DPI) delivering placebo to match the experimental drug. Participants received one dose of two inhalations.

SUMMARY:
The primary objective of this study is to evaluate the efficacy of a single dose (2 inhalations, 180 mcg total) of Albuterol SPIROMAX (90 mcg per inhalation) versus placebo in patients with EIB.

DETAILED DESCRIPTION:
This study is a single-dose, randomized, double-blind, placebo-controlled, 2-treatment, 2-sequence, 2-way crossover, multicenter study in patients with a documented history of EIB, with or without underlying asthma. Each patient will participate in the study for approximately 5 weeks. Each patient will complete 2 screening visits (SV1 and SV2), 2 treatment visits (TV1 and TV2), and a follow-up telephone call (FV).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent/assent: For patients 18 to 50 years of age, inclusive, written informed consent signed and dated by the patient before conducting any study related procedures and review of Health Insurance Portability and Accountability Act of 1996 (HIPAA) authorization; for patients 12 to 17 years of age, inclusive, written informed consent signed and dated by the parent/legal guardian and written assent signed and dated by the patient before conducting any study related procedure and review of HIPAA authorization.
* Male or female patients 12 to 50 years of age, inclusive, as of SV1.
* If female, is currently not pregnant, breastfeeding, or attempting to become pregnant, has a negative serum pregnancy test, and is of non-childbearing potential.
* Documented history of EIB, with or without underlying asthma. The underlying asthma must be well-controlled (in the investigator's judgment) as per the National Asthma Education and Prevention Program, Expert Panel Report (NAEPP, EPR-3).
* Other criteria apply.

Exclusion Criteria:

* Requires a rescue bronchodilator following the exercise challenge at SV1 for a decrease in FEV1 that does not return to within 20% of their pre-exercise challenge FEV1 within 30 minutes after administration of the rescue medication.
* Pregnant, nursing, or plans to become pregnant or donate gametes (ova or sperm) for in vitro fertilization during the study period or for 30 days after the patient's last study related visit (for eligible patients only-if applicable).
* Participation in any investigational drug trial within the 30 days preceding SV1 or planned participation in another investigational drug trial at any time during this trial.
* A known hypersensitivity to albuterol or any of the excipients in the formulation.
* History of severe milk protein allergy.
* History of a respiratory infection or disorder (including, but not limited to bronchitis, pneumonia, otitis media, acute or chronic sinusitis, influenza, etc) that has not resolved within the 2 weeks preceding SV1.
* Other criteria apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Teva Investigational Site 10557, San Diego, California
  - Teva Investigational Site 10555, Denver, Colorado
  - Teva Investigational Site 10558, Denver, Colorado
  - Teva Investigational Site 10559, Wheaton, Maryland
  - Teva Investigational Site 10560, North Dartmouth, Massachusetts
  - Teva Investigational Site 10556, Raleigh, North Carolina

REFERENCES:
- [Derived] Ostrom NK, Taveras H, Iverson H, Pearlman DS. Novel albuterol multidose dry powder inhaler in patients with exercise-induced bronchoconstriction: A single-dose, double-blind, randomized, 2-way crossover study. Respir Med. 2015 Nov;109(11):1410-5. doi: 10.1016/j.rmed.2015.09.004. Epub 2015 Sep 8. PMID 26475054

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 64 patients with EIB were screened. Of the 26 patients who did not participate in the study, 23 were excluded on the basis of inclusion/exclusion criteria, 2 patients withdrew consent, and 1 patient was withdrawn for other reason(s) before the baseline visit.
Period: Overall Study
Arm/Group | Albuterol Spiromax / Placebo Spiromax | Placebo Spiromax / Albuterol Spiromax
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Albuterol Spiromax / Placebo Spiromax | Placebo Spiromax / Albuterol Spiromax | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (7.11) | 31.9 (8.87) | 31.8 (7.93)
Age, Customized [Number; unit: participants]
  <18 years | 1 | 1 | 2
  >=18 years | 18 | 18 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 10 | 9 | 19
Race/Ethnicity, Customized [Number; unit: participants]
  White | 14 | 16 | 30
  Black | 4 | 2 | 6
  Asian | 0 | 1 | 1
  Other | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 2 | 2 | 4
  Non-Hispanic and non-Latino | 17 | 17 | 34
Weight [Mean (Standard Deviation); unit: kg] | 82.7 (15.54) | 74.2 (21.04) | 78.4 (18.75)
Height [Mean (Standard Deviation); unit: cm] | 171.4 (12.06) | 169.8 (11.46) | 170.6 (11.63)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.1 (4.00) | 25.3 (4.58) | 26.7 (4.47)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Percentage Fall From Baseline in Forced Expiratory Volume in 1 Second (FEV1) up to 60 Minutes After the Exercise Challenge
Description: A centralized spirometry data collection system was used to reduce FEV1 variability between and within patients and between each participating study center.
  The percentage fall was defined as 100*(baseline-post baseline)/baseline. The baseline FEV1 is the test day FEV1 measured 5 minutes before the exercise challenge (30 minutes postdose). FEV1 post exercise challenge were measured 5 (±5), 10 (±5), 15 (±5), 30 (±5), and 60 (±10) minutes after completion of the exercise challenge.
  The exercise challenge consisted of the participant running on a motor-driven treadmill (with adjustable speed and incline). The treadmill was set at a speed and incline sufficient to increase the participant's heart rate to ≥80% of the maximum rate for age (220 bpm-age in years) for a period of either 6, 7, or 8 minutes using a stepped-exercise protocol in accordance with ATS guidelines (American Thoracic Society 2000). Conditions were repeated for subsequent challenges.
Time Frame: Days 1 and 7; up to 60 minutes post-exercise challenge
Population: Full analysis set
Measure: Mean (Standard Error); unit: percentage change from baseline FEV1
Groups:
- Albuterol Spiromax 180 mcg: Single dose of Albuterol Spiromax, 180 mcg (2 inhalations of 90 mcg/inhalation)
- Placebo Spiromax: Single dose of Placebo Spiromax (2 inhalations)
Arm/Group | Albuterol Spiromax 180 mcg | Placebo Spiromax
Number analyzed (Participants) | 38 | 38
percentage change from baseline FEV1 | 6.21 (1.443) | 22.38 (1.444)
Statistical Analysis 1: Comparison: Albuterol Spiromax 180 mcg vs Placebo Spiromax; Test type: Superiority or Other; p < 0.0001, mixed-effect analysis of covariance — Significance level is 0.05; Fixed effects of sequence, trt group, period, and center, within period baseline FEV1 as a covariate, and random effect for patient within sequence; Mean Difference (Final Values) = -16.2, 95% CI 2-sided [-20.19 to -12.14], Standard Error of Mean 1.982

2. Secondary Outcome: Percentage of Participants Whose Maximum Percentage Decrease From the Baseline Forced Expiratory Volume in 1 Second (FEV1) Post-Exercise Challenge Was <10%
Description: Participants were classified as protected if the maximum percentage decrease from baseline FEV1 after exercise was less than 10%. Data represents the percentage of participants who were classified as protected.
Time Frame: Days 1 and 7; up to 60 minutes post-exercise challenge
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Albuterol Spiromax 180 mcg | Placebo Spiromax
Number analyzed (Participants) | 38 | 38
percentage of participants | 84.21 | 15.79
Statistical Analysis 1: Comparison: Albuterol Spiromax 180 mcg vs Placebo Spiromax; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Terms for treatment and period, computed with the generalized estimating equations (GEE) algorithm, which adjusts for potential correlation between measurements on the same patient. Significance level of 0.05; Mean Difference (Final Values) = 0.68, 95% CI 2-sided [0.53 to 0.84], Standard Error of Mean 0.075

3. Secondary Outcome: Participants Whose Maximum Percentage Decrease From the Baseline Forced Expiratory Volume in 1 Second (FEV1) Post-Exercise Challenge Was >20%
Description: Participants were classified as unprotected if the maximum percentage decrease from baseline FEV1 after exercise was more than 20%. Data represents the number of participants who were classified as unprotected.
Time Frame: Days 1 and 7; up to 60 minutes post-exercise challenge
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Albuterol Spiromax 180 mcg | Placebo Spiromax
Number analyzed (Participants) | 38 | 38
participants | 1 | 22

ADVERSE EVENTS:
Time Frame: Days 1-14
Arm/Group | Albuterol Spiromax 180 mcg | Placebo Spiromax
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.